CLINICAL TRIAL: NCT04790149
Title: Synergistic Effect of tDCS and Neuromotor Recruitment on Functional Recovery in Chronic Paraplegia: A Randomized Controlled Trial
Brief Title: Effectiveness of NEUROM and tDCS for Motor Recovery in Chronic Paraplegia
Acronym: NEUROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Ahmad Rifai Sarraj, Professor, Lebanese University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE-EDST-10-2019
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Neurorehabilitation; Motor and Sensory Recovery; Physical Therapy
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Physical Therapy Modalities; Transcranial Direct Current Stimulation; NeuroM protein, chicken

STUDY DESIGN:
Intervention Model Description: 3 groups receiving parallel different interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Group (Sham Comparator): Conventional usual Rehabilitation is administered to a group of patients without any effect on their recovery
  Interventions: Other: Conventional Rehabilitation
- NEUROM (Experimental): participants received the new protocol of a method called NEUROM consisting of 3 phases of treatment : Motor Imagery training, active rehabilitation and functional rehabilitation
  Interventions: Other: NEUROM
- NEUROM combined with tDCS (Experimental): same as the second arm of NEUROM combined with transcranial direct stimulation
  Interventions: Other: NEUROM + tDCS

INTERVENTIONS:
Other: Conventional Rehabilitation — Motor Imagery Training combined with Active functional exercises
  Other Names: Physical Therapy
  Arms: Conventional Group
Other: NEUROM + tDCS — NEUROM combined to tDCS
  Arms: NEUROM combined with tDCS
Other: NEUROM — protocol to induce motor recovery
  Arms: NEUROM

SUMMARY:
Traumatic Spinal Cord Injury (TSCI) is a catastrophic, unexpected, and devastating event that can occur along the spinal column (cervical, thoracic, and lumbar). Traditional views describe the spinal cord as a protected bundle of nerves connecting the brain to the body. TSCI often results in life-threatening conditions including varying degrees of motor paralysis, sensory loss, and impairment of bowel, bladder, sexual, and other physiologic functions.

In this study, the investigators propose a new experimental rehabilitative protocol for TSCI patients called the Neural Motor Recruitment Method (NEUROM). This method is based on histological and functional reorganization models following TSCI, Motor Imagery (MI) concepts, and targeted sensory inputs related to motor recovery. It is hypothesized that this new method can enhance sparing-induced plasticity and increase motor and sensory recovery in SCI patients, especially when combined with Transcranial Direct Current Stimulation (tDCS).

DETAILED DESCRIPTION:
PARTICIPANTS Fifty participants with paraplegia will be recruited from inpatient rehabilitation hospitals. Patients will be treated at Rahma Hospital for Rehabilitation in Tripoli and the Physical Therapy Center of the Faculty of Public Health-I in Hadath.

INCLUSION/EXCLUSION CRITERIA Main inclusion criteria include: age between 18-45 years; diagnosis of chronic spinal cord injury (defined as at least 3 months post-injury); and injury level below T10 with an American Spinal Injury Association Impairment Scale (AIS) classification of A, B, or C. Ethical committee approval will be obtained from the Lebanese University official ethical committee, and informed consent will be obtained from all participants in accordance with the Declaration of Helsinki.

Exclusion criteria include: neuropsychiatric comorbidities; traumatic brain injury (TBI); involvement in any specific program of rehabilitation other than the conventional protocol since injury; and contraindications to tDCS (such as metal in the head or implanted medical devices). Patients with a history of seizure, use of medications containing sodium channel blockers (e.g., carbamazepine), or any substance abuse will be excluded. Patients with severe spasticity (greater than or equal to 3 out of 4 on the Modified Ashworth Scale) will also be excluded.

Prior to the experiment, patients must have received conventional physiotherapy and demonstrated stable lower limb functional scores; performance must not change from the end of conventional therapy until the first baseline measurements.

STUDY DESIGN & ARMS All subjects will be randomly assigned into three groups:

Reference Group (n=10): Participants will receive a standardized conventional intervention (stretching, strengthening, neuro-muscular facilitation).

NEUROM Group (n=20): Participants will receive the Neural Motor Recruitment Method (NEUROM).

NEUROM + tDCS Group (n=20): Participants will receive the NEUROM protocol combined with tDCS.

All participants will undergo a detailed medical examination, with particular attention to the experimental group receiving tDCS to eliminate adverse effects. Before every session, participants will be prepared for the closed-loop rehabilitation protocol by 20 minutes of static stretching of the lower legs, specifically the hamstrings and soleus muscles.

INTERVENTIONS

Conventional Rehabilitation Program: The conventional control group will undergo therapeutic exercises including: repetitive neuromuscular facilitation, passive and active mobilization, strengthening, endurance exercises, and musculoskeletal interventions (static and dynamic stretching).

Neural Motor Recruitment (NEUROM): Patients in the NEUROM and NEUROM+tDCS groups will receive daily home Motor Imagery (MI) training with 20 minutes of stretching for 10 days. MI training will be individually delivered in a quiet room designed for this purpose. Participants will lay on a bed facing a 43-inch screen located 3.5 meters away, with the center of the screen 1.2 meters from the floor. The screen will display a 5-minute video of two feet repeating large movements of dorsi- and plantar flexion. Instructions will be detailed and read aloud. An audio output will guide the subject to feel the movement (kinesthetic imagery) with the instruction: "Imagine yourself performing the feet movement without actually executing it with your eyes closed."

Transcranial Direct Current Stimulation (tDCS): The combined group will receive NEUROM + tDCS. The StarstimNE non-invasive wireless tDCS neurostimulator (Neuroelectrics®, Barcelona, Spain) will be used. A wireless neoprene cap based on the International 10-20 System will be placed on the participant's head by aligning the central Cz electrode position with the vertex. Small Ag/AgCl gelled electrodes (3.14 cm²) will be used. In all sessions, one electrode will be placed on the left M1 and the other on the right M1 (corresponding to C3 and C4). The montage will alternate: in one session the anode will be on the left M1 and the cathode on the right M1 (AL-CR), and in the next session, the polarity will be reversed (AR-CL). DC current will be increased over 7 seconds to 1 mA and maintained for 20 minutes. During tDCS, the participant will be asked to perform kinesthetic imagery.

OUTCOME MEASURES

Vividness of Motor Imagery Questionnaire (VMIQ): Participants will indicate the vividness of an imagined movement on a 5-point scale (1: excellent/lively as actual performance; 5: no image at all).

Assessment of Movement Attempt (AMA) and Execution: The motor task consists of repetitive alternating dorsal and plantar flexion of the right foot (30°-0°-45°) at a self-paced rhythm. The perceived intensity and frequency of attempted movements will be rated in a structured interview. Answers are noted as qualitative descriptors and rated on a 6-point scale (1: very weak/rare; 6: very high/often).

ASIA Examinations: Motor and sensory examinations will be performed by SCI-experienced physical therapists at baseline, week 1, week 2, and week 4. Five key muscle groups will be assessed (total score /50) and sensation will be recorded for 12 key sensory points (Light Touch and Pin Prick; max score /48).

Visual Analog Scale (VAS): Used to measure introspective perception of movement during the illusion condition. Participants will rate the strength of the kinesthetic illusion from 0 mm (no sensation) to 100 mm (feels exactly like actual movement).

EXPECTED OUTCOMES & APPLICABILITY Priming the motor cortex to augment functional benefits with peripheral training is a relatively new approach. Research is needed to increase the effectiveness of physical rehabilitation in Spinal Cord Injury. The investigators anticipate that distinguishing between therapies with unequal impacts on outcomes will answer clinical questions regarding non-conventional strategies. The findings may support the hypothesis that modulating excitatory input of the corticospinal tracts combined with motor imagery in a closed-loop protocol is a promising strategy for improving lower limb functions in chronic paraplegia.

ELIGIBILITY:
Inclusion Criteria

* Age: Between 16 and 45 years.
* Diagnosis: Chronic spinal cord injury (at least 3 months post-injury).
* Level of Injury: Lower dorsal (below T10) or lumbar.
* Classification: American Spinal Injury Association Impairment Scale (AIS) grade A, B, or C.
* Signed Informed Consent.

Exclusion Criteria

* Comorbidities: Neuropsychiatric comorbidities or Traumatic Brain Injury (TBI).
* Concurrent Treatment: Involvement in any specific rehabilitation program other than the conventional protocol since injury.
* tDCS Contraindications: Presence of metal in the head or implanted medical devices (e.g., pacemaker, cochlear implant).
* Seizure History: Any history of epilepsy or seizures.
* Medications: Current use of medications containing sodium channel blockers (e.g., carbamazepine) or history of substance abuse.
* Spasticity: Severe spasticity defined as a Modified Ashworth Scale score ≥ 3.

Crucial Data Fixes (You must update these fields in the registry UI):

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Lower Extremity Motor Score (LEMS) according to ISNCSCI Standards | Baseline and Week 3 (End of Intervention)
  Motor function is assessed using the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI). Five key muscles in each lower limb (L2-S1) are graded on a scale of 0 (total paralysis) to 5 (normal active movement). The total score ranges from a minimum of 0 to a maximum of 50. Higher scores indicate better motor function.
Change in Sensory Scores (Light Touch and Pin Prick) | Baseline and Week 3
  Sensation is evaluated at 12 key sensory points on both lower limbs according to ISNCSCI standards. Each point is graded as 0 (absent), 1 (impaired), or 2 (normal).
  Light Touch Total Score Range: 0 to 48. Pin Prick Total Score Range: 0 to 48. Higher scores indicate better sensory function.
Change in Assessment of Movement Attempt (AMA) Scores | Baseline and Week 3
  The AMA evaluates the patient's subjective ability to voluntarily attempt movement in the paralyzed limb. It consists of two sub-scales assessed during a structured interview:
  Intensity of Motor Attempt: Rated on a 6-point scale ranging from 1 (very weak feeling) to 6 (very high intensity).
  Frequency of Spontaneous Attempt: Rated on a 6-point scale ranging from 1 (very rare) to 6 (very often/daily). Scores are reported individually for each sub-scale. Higher scores indicate better volitional drive and motor intent.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Rifai Sarraj, PhD, Principal Investigator — Lebanese University
Locations (1):
- Lebanese University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No